CLINICAL TRIAL: NCT04469959
Title: Dopaminergic Dysfunction in Late-Life Depression
Acronym: D3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Emory University (Other); University of Pittsburgh (Other); University of Pittsburgh Medical Center (Other); Rutgers University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Warren Taylor, Professor of Psychiatry, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201172
Record Dates: First submitted 2020-07-02; First posted 2020-07-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Late Life Depression; Cognitive Decline; Depressive Disorder, Treatment-Resistant; Levodopa; Gait Impairment
Keywords: Antiparkinson agent; Levodopa; Elderly; Depressive Disorder, major
MeSH Terms: conditions — Cognitive Dysfunction; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Levodopa; Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-Dopa First / Placebo Second (Experimental): STEP 1(3 weeks): Participants initially assigned to L-DOPA will begin with a Week 1 L-DOPA daily dosage of 150mg, (1.5 25mg carbidopa/100mg levodopa capsules) at 9am. Week 2 will increase to a L-DOPA daily dose of 300mg (1.5 25mg carbidopa/100mg levodopa capsules) at 9am and 5pm, followed by a Week 3 L-DOPA daily dose of 450mg (1.5 25mg carbidopa/100mg levodopa capsules) three times daily. After completing post-trial assessments, participants then enter a 1 week taper period before proceeding to Step 2.
  Step 2 (3 Weeks): Participants will receive matching placebo capsules daily. Participants take placebo capusles once daily during week 1 (9am), twice daily during week 2 (9am, 5pm), and three times daily during week 3 (9am, 1pm, 5pm) over three weeks. Following post-trial assessments, participants then enter a 1-week taper period and study drug is withdrawn.
  Interventions: Drug: L-Dopa; Drug: Placebo
- Placebo First / L-Dopa Second (Placebo Comparator): Step 1 (3 Weeks): Participants will receive matching placebo capsules daily. Participants take placebo capsules once daily during week 1 (9am), twice daily during week 2 (9am, 5pm), and three times daily during week 3 (9am, 1pm, 5pm) over three weeks. Following post-trial assessments, participants then enter a 1-week taper period before proceeding to Step 2.
  Step 2 (3 Weeks): Participants will begin with a Week 1 L-DOPA daily dosage of 150mg, (1.5 25mg carbidopa/100mg levodopa capsules) at 9am. Week 2 will increase to a L-DOPA daily dose of 300mg (1.5 25mg carbidopa/100mg levodopa capsules) at 9am and 5pm, followed by a Week 3 L-DOPA daily dose of 450mg (1.5 25mg carbidopa/100mg levodopa capsules) three times daily. After completing post-trial assessments, participants then enter a 1 week taper period and study drug will be discontinued.
  Interventions: Drug: L-Dopa; Drug: Placebo

INTERVENTIONS:
Drug: L-Dopa — Generic 25/100mg carbidopa/levodopa (Sinemet)capsules will be administered in this study. Participants will begin randomized double blinded 3- week trial of Levodopa. Dose titration starting at 150 mg /daily to maximum of 450 mg daily three times a day for three weeks.
  After one week of taper participants will enter step 2 phase of study where carbidopa/levodopa matched placebo will be administered for 3 weeks afterwards dose will be slowly tapered over next 7 days.
  Other Names: carbidopa/levodopa (Sinemet); 25/100 placebo capsules
Drug: Placebo — Step 1 (3 weeks) Carbidopa/levodopa-matched placebo capsules 3 times. Followed by 1 week of taper. Step2(3 weeks):150-450mg carbidopa/levodopa 3 times daily for three weeks .Followed by 1 week of taper.
  Other Names: 25/100 placebo capsules

SUMMARY:
Late-Life Depression (LLD), or depression in older adults, often presents with motivational deficits, deficits in performance in cognitive domains including processing speed and executive dysfunction, and mobility impairments. This triad of findings implicate dopaminergic dysfunction as a core pathophysiologic feature in depression, and may contribute to cognitive decline and motor disability. Normal aging results in brain-wide dopamine declines, decreased D1/D2 receptor density, and loss of dopamine transporters. Although brain changes associated with depression and aging converge on dopamine circuits, the specific disturbances in LLD and how responsive the system is to modulation remain unclear. In this study, investigators are testing integrative model that aging, in concert with pro-inflammatory shifts, decreases dopamine signaling. These signally changes affects behaviors supported by these circuits, in the context of age-associated cortical atrophy and ischemic microvascular changes, resulting in variable LLD phenotypes. Investigators propose a primary pathway where dopaminergic dysfunction in depressed elders contributes to slowed processing speed and mobility impairments that increase the effort cost associated with voluntary behavior. The central hypothesis of this study is that late-life depression is characterized by dysfunction in the dopamine system and, by enhancing dopamine functioning in the brain. By improving cognitive and motor slowing, administration of carbidopa/levodopa (L-DOPA) will improve depressive symptoms.

DETAILED DESCRIPTION:
Late Life Depression (LLD) is a prevalent, disabling, and at times lethal condition for which currently available treatments are often ineffective. No prior study has comprehensively examined dopamine-dependent behaviors (i.e., reward processing, cognition, motor function) in LLD, and none has integrated positron emission tomography (PET), multimodal magnetic resonance imaging (MRI), neuropsychological evaluation, and mobility assessments. Should cognitive and motor slowing result in altered effort-based decision making as researchers hypothesize, treatment development may shift from addressing mood and hedonic responses toward facilitating cognition and movement, reducing the effort cost of voluntary behavior, and promoting behavioral activation.

This study, across collaborative sites, will enroll 100 evaluable elderly depressed outpatients who enter baseline study procedures and who exhibit evidence of dopaminergic dysfunction, characterized as either slowed processing speed or slowed gait speed. To disentangle depression effects from age-related changes, 70 never-depressed elders also will complete baseline evaluation. To achieve this goal, at Vanderbilt University Medical Center (VUMC) the investigators will enroll 80 depressed elders and 50 never-depressed elders who complete baseline study procedures. The University of Pittsburgh Medical Center will enroll an additional 20 depressed elders and 20 never-depressed elders who complete baseline study procedures.

Assessments include PET imaging of receptor density, neuromelanin-sensitive MRI (NM-MRI) measurement of nigrostriatal status, task-based MRI focused on effort-based decision making and reward processing, and comprehensive psychiatric, neurocognitive, and physical performance evaluation. Depressed participants then will be randomized to levodopa (L-DOPA) or placebo for 3 weeks, followed by repeat multimodal MRI and cognitive/behavioral assessments. In a cross-over phase, participants will receive the opposite intervention for an additional 3 weeks followed by clinical and cognitive assessments only. This mechanistic probe allows the investigators to examine the contributions and interrelationships of dopamine-dependent processes in LLD and evaluate the responsivity of dopamine systems in LLD to pharmacological stimulation.

AIM 1: To characterize dopaminergic dysfunction in LLD at molecular, circuit, and behavioral levels.

Hyp 1: Compared to age- and gender-matched controls on baseline functional MRI (fMRI), LLD participants will be less willing to expend effort for rewards and exhibit lower prefrontal cortex and striatal activation on the Effort Expenditure for Rewards Task (EEfRT). Hyp 2: Across all participants, lower striatal [18F]-FDOPA relative influx rate, lower midbrain & striatal [18F]-fallypride binding, and lower NM-MRI signal in the substantia nigra, pars compacta will predict lower performance across RDoC domains: Positive Valence (impaired willingness to expend effort, decreased neural activations on the EEfRT), Cognitive (slowed processing speed and executive dysfunction), and Sensorimotor (slowed gait speed). Hyp 3: Across all participants, slowed processing and gait speed likewise will predict lower willingness to expend effort on the EEfRT.

AIM 2: To examine responsivity of dopamine circuits in LLD to stimulation with L-DOPA.

Hyp 1: Compared to placebo, L-DOPA will result in greater normalization of neural activations and improved behavioral performance in Positive Valence, Cognitive, and Sensorimotor domains. Hyp 2: Baseline PET and NM-MRI measures will moderate L-DOPA effects. The greatest improvements will be observed in those with the lowest baseline [18F]-FDOPA relative influx rate, [18F]-fallypride binding, and NM-MRI signal.

Exploratory Aims: 1) To investigate associations of baseline proinflammatory markers with dopaminergic function across molecular, circuit, cognitive and behavioral levels of analysis. 2) To evaluate the durability of L-DOPA effects on RDoC domains in the crossover phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years
2. Diagnostic and Statistical Manual-5 (DSM5) diagnosis of Major Depressive Disorder, Persistent Depressive Disorder, or Depression Not Otherwise Specified (NOS)
3. MADRS score ≥ 15
4. Decreased processing speed (0.5 SD below age-adjusted norms on the WAIS-IV Coding task or Trail Making Test, Part A) or decreased motor speed (gait speed/average walking speed on 15' course ≤ 1m/s, or 0.5 SD below age-, gender- and education-adjusted norms on the grooved pegboard test)
5. Capable of providing informed consent and adhering to study procedures

Exclusion Criteria:

1. Diagnosis of substance abuse or dependence (excluding Tobacco Use Disorder) in the past 12 months
2. Other psychiatric disorders including a history of psychosis, psychotic disorder, mania, or bipolar disorder. Other comorbid psychiatric disorders are allowable if the depressive disorder diagnosis is considered to be the primary problem
3. Primary neurological disorder, including dementia, stroke, Parkinson's disease, epilepsy, etc
4. SBT > 10
5. MADRS suicide item > 4 or other indication of acute suicidality
6. History of inpatient psychiatric hospitalization in the last year;
7. History of suicidal ideation in the last 6 months, operationalized as a 'yes' response to item 4 or 5 in the "Suicidal Ideation" section of the Columbia-Suicide Severity Rating Scale (CSSRS)
8. Any suicidal behavior in the last year (operationalized as a 'yes' response to any item in the "Suicidal Behavior" section of the CSSRS, including actual interrupted, aborted, or preparatory acts)
9. Current or recent (within the past 2 weeks) treatment with antipsychotics or mood stabilizers, or use of antidepressants where washout is not advisable
10. History of hypersensitivity, allergy, or intolerance to Carbidopa/levodopa
11. Any physical or intellectual disability adversely affecting ability to complete assessments
12. Unstable medical illness
13. Mobility limiting osteoarthritis of any lower extremity joints, symptomatic lumbar spine disease, or history of joint replacement / spine surgery that limits mobility
14. Diagnosis of HIV
15. History of significant radioactivity exposure (nuclear medicine studies or occupational exposure).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in WAIS-R Digit Symbol Task Score | Baseline, after week 3, and after week 6
  Wechsler Adult Intelligence Scale(WAIS-R) Digit Symbol Task score will be used to measure processing speed. A composite score is derived with two other test scores of WAIS-R Pattern Comparison Test Score by extracting latent fact and factor loadings, creating a purer measure of processing speed. Higher scores indicate better performance.
Change in Pattern Comparison Test Score | Baseline, after week 3, and after week 6
  Pattern Comparison Test score will be used to measure processing speed. A composite score is derived with two other test scores of WAIS-R by extracting latent fact and factor loadings, creating a purer measure of processing speed. Higher scores indicate better performance.
Change in Letter Comparison Test Score | Baseline, after week 3, and after week 6
  Letter Comparison Test score will be used to measure the processing speed. A composite score is derived with two other test scores of WAIS-R by extracting latent fact and factor loadings, creating a purer measure of processing speed. Higher scores indicate better performance.
Change in NIH EXAMINER Test Score | Baseline, after week 3, and after week 6
  This neuropsychological test battery assesses a range of executive functions. Tasks measuring working memory, inhibition, set shifting, fluency, insight, and planning and 3 self-report questionnaires rating social cognition and behavior. Higher scores indicate better performance.
Change in Gait pattern | Baseline, after week 3, and after week 6
  Gait will be assessed with a single and dual task (ST, DT) using the GaitRite system (VUMC) or Zeno walkway system (UPMC), which assesses gait parameters in real time (gait speed, cadence, stride length). Changes in these parameters will reflect changes in gait slowness.
Change in Effort Expenditure for Rewards Task (EEfRT) | Baseline to after week 3
  In this functional Magnetic Resonance Imaging task, participants decide whether to work harder for a larger reward (high number of finger presses with their pinky) or expend less energy (low number of presses with a dominant index finger) for a lesser reward, with lower rewards being $1 dollar and higher rewards ranging from $1.20 to $5. Participants receive information about the probability of winning on each trial regardless of their pick and one trial from each run is randomly picked for payout. The primary outputs on this task are the percentage of time participants choose the high cost / high reward option on the EEfRT and associated neural activation patterns in prefrontal cortex (PFC) and striatum.

SECONDARY OUTCOMES:
Change in NIH Toolbox Cognition Battery Scores | Baseline, after week 3, and after week 6
  This is a brief and psychometrically sound set of 7 computerized instruments providing an overall cognitive index from measures of 6 cognitive domains.
Monetary Incentive Delay Task | Baseline and after week 3
  This functional Magnetic Resonance Imaging task assesses neural response during reward anticipation and receipt. On each trial, participants are presented with a 2000msec cue indicating that trial's reward value ($0, $1, or $5). After the cue, a 2000-2500 msec delay period ensues as the participant waits for the target. Participants press a button as quickly as possible when the target is visible. After another delay lasting from 950 to 2800 msec, a feedback screen lasting 2500msec appears indicating the outcome ("Hit!" or "Miss!") for each trial, with a brief interval before the next trial. the primary contrast for analyses is the contrast of Cue $5 - Cue $0 to brain activation during reward anticipation. The contrast of Hit vs. Miss on both $5 and $1 trials is the primary index of reward receipt.
Change in MADRS (Montgomery Asberg Depression Rating Scale) Score | Baseline and weekly thereafter for 6 weeks
  Secondary outcome measured by the total score of the clinician rated MADRS, a measure of depression severity. The MADRS total score range is 0-60, where higher scores indicate greater depression severity.
Change in QIDS (Quick Inventory of Depressive Symptomatology) Score | Baseline and weekly thereafter for 6 weeks
  QIDS-16-item, a participant-rated measure of depressive symptomatology. The total score ranges from 0 to 27, with higher scores indicative of greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Taylor, MD,MHSc, Study Director — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt Psychiatric Hospital, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
This study will include clinical, cognitive, and neuroimaging data from older depressed subjects. The final dataset will include clinical information about subject psychiatric diagnoses, psychiatric and medical history, cognitive data, and response to L-dopa . The investigators will share data via the National Database for Clinical Trials related to Mental Illness (NDCT). NDCT provides a secure platform for data-sharing allowing for communication of research data, tools, and supporting documents. As required by NDCT, the investigators will obtain a Global Unique Identifier (GUID) for each participant. The investigators will additionally follow NDCT requirements to certify and review data, as well as timeline requirements for data submission and data sharing. Sharing of neuroimaging data will also be facilitated by an XNAT system (xnat.org). XNAT is an open-source informatics software platform that assists in the management and archiving of imaging data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared according to policies from the NDCT and NDA (NIMH Data Archive). Descriptive data, outcome measures and analyzed data will be shared will be shared within 4 months of when a publication is accepted. Study data will be shared through the NDCT indefinitely.
Access Criteria: The NIH will provide access to scientific investigators for research purposes. Qualified researchers who have completed a Data Use Certification and received approval from the NDA Data Access Committee (DAC) may be approved to access broadly shared data. A separate request process exists for access to data in federated sources. Additionally, the DAC and support staff at NIH have access to NDA shared data.
URL: https://nda.nih.gov

REFERENCES:
- [Background] Taylor WD. Clinical practice. Depression in the elderly. N Engl J Med. 2014 Sep 25;371(13):1228-36. doi: 10.1056/NEJMcp1402180. No abstract available. PMID 25251617
- [Background] Treadway MT, Bossaller NA, Shelton RC, Zald DH. Effort-based decision-making in major depressive disorder: a translational model of motivational anhedonia. J Abnorm Psychol. 2012 Aug;121(3):553-8. doi: 10.1037/a0028813. Epub 2012 Jul 9. PMID 22775583
- [Background] Kunisato Y, Okamoto Y, Ueda K, Onoda K, Okada G, Yoshimura S, Suzuki S, Samejima K, Yamawaki S. Effects of depression on reward-based decision making and variability of action in probabilistic learning. J Behav Ther Exp Psychiatry. 2012 Dec;43(4):1088-94. doi: 10.1016/j.jbtep.2012.05.007. Epub 2012 May 31. PMID 22721601